CLINICAL TRIAL: NCT01576770
Title: In Children, Does the Use of Synera Patch for Local Analgesia Before Vascular Access Reduce Pain Associated With Propofol Injection for Anesthesia Induction?
Brief Title: In Children, Does Using a Synera Patch Decrease Pain When Injecting Propofol at Anesthesia Induction?
Acronym: Synera patch
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: ZARS Pharma Inc. (Industry)
Responsible Party: Principal Investigator, Samia Khalil, Professor of Pediatric Anesthesia, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-12-0042
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Pain on Propofol IV Injection
Keywords: propofol; Pain; Synera Patch; Gebauer's Ethyl Chloride topical anesthetic
MeSH Terms: conditions — Pain | interventions — Ethyl Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ethyl chloride vapocoolant spray (Active Comparator): Half of the patients will randomly be assigned to receive Gebauer's ethyl choride topical anesthetic vapo-coolant spray immediately prior to placing a 22 gauge intravenous catheter.
  Pain in this group will be evaluated at the time of IV placement by an independent observer (unblinded) and the patient on a 0-10 scale. Pain will again be evaluated when propofol is injected at anesthesia induction by a blinded observer and the staff anesthesiologist (also blinded) on a scale of 1-4.
  Blinding will occur following IV placement by draping and securing the hand and IV site with Coban self-adherent elastic wrap to cover any skin changes due to the ethyl chloride or the patch.
  Interventions: Drug: Gebauer's Ethyl Chloride
- Synera Patch (Experimental): The other half of the patients will randomly be assigned to receive Synera Patches, to be applied to the dorsum of both hands, at least 30 minutes before placing a 22 gauge intravenous catheter.
  Pain in this group will be evaluated at the time of IV placement by an independent observer (unblinded) and the patient on a 0-10 scale. Pain will again be evaluated when propofol is injected at anesthesia induction by a blinded observer and the staff anesthesiologist (also blinded) on a scale of 1-4.
  Blinding will occur following IV placement by draping and securing the hand and IV site with Coban self-adherent elastic wrap to cover any skin changes due to the patch or ethyl chloride.
  Interventions: Device: lidocaine/tetracaine transdermal patch (NDC 43469-864-01)

INTERVENTIONS:
Device: lidocaine/tetracaine transdermal patch (NDC 43469-864-01) — 70 mg lidocaine / 70 mg tetracaine
  Other Names: NDC 43469-864-01
  Arms: Synera Patch
Drug: Gebauer's Ethyl Chloride — Spray is to be applied topically to skin (dorsum of the hand for study purposes)until it turns white or for up to 10 seconds.
  Other Names: CHLOROETHANE, HYDROCHLORIC ETHER; NDC 45951-0123
  Arms: ethyl chloride vapocoolant spray

SUMMARY:
The purpose of this study is to evaluate if the Synera Patch (lidocaine/tetracaine patch), used to numb the skin before IV placement, is effective in reducing pain associated with propofol IV administration when inducing general anesthesia, compared to Gebauer's Ethyl Chloride topical anesthetic skin refrigerant.

DETAILED DESCRIPTION:
Commonly, anesthesiologists inject Propofol, a sleeping medication, intravenously to induce general anesthesia. Propofol injection is associated with pain that can be severe.

The investigators also place a lidocaine/tetracaine skin patch (Synera) to decrease pain associated with IV placement. Because the local anesthetics of the Synera patch diffuse deep underneath the skin, in this study the investigators would like to evaluate whether the application of Synera Patch can decrease the pain associated with propofol injection.

Children will be randomized to receive either the patch or the Ethyl Chloride before the IV placement. A total of 33 patients will be enrolled in each group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, outpatient children, 6-17 years old
* American Society of Anesthesiologist Physical Classification rating of 1 or 2
* Elective procedure requiring general anesthesia at Memorial Herman Hospital, The Medical Center, Houston, Texas

Exclusion Criteria:

* Skin disease or infection (on dorsum of hands)
* Allergy to lidocaine or tetracaine

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-10 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Number of children in each group who do not feel pain or have mild pain on propofol injection. | Within one hour, plus or minus one half hour
  The primary outcome variable is the success/failure of therapy. The therapy is considered a success if a child feels no pain OR has mild pain.

SECONDARY OUTCOMES:
Pain intensity | Within one hour, plus or minus one half hour
  A blinded independent observer and a blinded anesthesiologist will rate pain on propofol injection according to a pain scale:
  1. - no pain
  2. - mild pain (associated with facial expression of pain)
  3. - moderate pain (pulling/withdrawal of the arm)
  4. - severe pain (screaming)

CONTACTS AND LOCATIONS:
Overall Officials: Samia N Khalil, M.D., Principal Investigator — University of Texas Health Sciences Center at Houston
Locations (1):
- Memorial Herman Hospital, Houston, Texas, United States